CLINICAL TRIAL: NCT01487668
Title: Life Goals Collaborative Care to Improve Health Outcomes in Mental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 10-340
Record Dates: First submitted 2011-11-21; First posted 2011-12-07 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Bipolar Disorder; Schizophrenia; Major Depressive Disorder; Schizoaffective Disorder; Cardiovascular Disease Risk
Keywords: chronic mental disorders; cardiovascular disease; behavior change
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Depressive Disorder, Major; Psychotic Disorders; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 - Usual Care (No Intervention): Usual care will include standard mental health and medical care available in the VA clinics but with no active management by the LGCC health specialist.
- Arm 2 - Life Goals Collaborative Care (Experimental)
  Interventions: Behavioral: Life Goals Collaborative Care

INTERVENTIONS:
Behavioral: Life Goals Collaborative Care — LGCC consists of 1) 10 self-management sessions that cover personal goal-setting and mental health symptom management reinforced through healthy lifestyles; 2) medical care management that includes identification of patient medical risk factors, monitoring of patient symptoms and medical needs via a registry over time; and 3) support for provider guidelines and community linkages.
  Arms: Arm 2 - Life Goals Collaborative Care

SUMMARY:
Persons with serious mental illness (SMI) are at increased risk of cardiovascular disease (CVD). The goals of this study are to test a treatment, Life Goals Collaborative Care to help promote health behavior change and improve mental health and physical health-related quality of life, as well as to get feedback from patients and providers on what is needed to help better coordinate the physical and mental health care of these patients.

DETAILED DESCRIPTION:
Background: VA patients with serious mental illnesses (SMI- e.g., schizophrenia, bipolar disorder) die an average of 13-18 years earlier compared to the general U.S. population, mostly from cardiovascular disease (CVD). Increased risk of CVD and related risk factors in persons with SMI is attributed to patient, provider, and system-level barriers including unhealthy behaviors exacerbated by mental health-related symptoms and barriers to access and continuity of care between physical and mental health services.

Objectives: The primary aim of this randomized controlled effectiveness trial (RCT) is to determine whether VA patients with SMI receiving Life Goals Collaborative Care (LGCC), a program that combines customized behavioral change strategies with chronic care management for SMI will experience, within 12 months: a) improved medical outcomes (e.g., reduced CVD risk factors, improved physical health-related quality of life), b) improved mental health outcomes, including reduced psychiatric symptoms or improved mental health-related quality of life or c) improved health behaviors, compared to VA patients with SMI receiving enhanced treatment as usual (i.e., dissemination of health behavior change materials in addition to standard VA medical and psychiatric care). Secondary aims that will inform further implementation of LGCC will be to assess utilization and cost differences of LGCC versus treatment as usual, determine the patient factors associated with LGCC treatment response, and identify the organizational factors associated with LGCC implementation.

Methods: LGCC is a groundbreaking psychosocial and behavior change intervention that is based on the Chronic Care Model (CCM) and consists of 1) 10 self-management sessions that cover personal goal-setting and mental health symptom management reinforced through healthy lifestyles; 2) medical care management that includes identification of patient medical risk factors, monitoring of patient symptoms and medical needs via a registry over time; and 3) support for provider guidelines and community linkages. The investigators will enroll individuals diagnosed with SMI and a CVD risk factor who are receiving care within the VA Ann Arbor Healthcare System mental health clinic, and who will be randomized to receive LGCC or enhanced treatment as usual. Key outcomes include changes in CVD risk factors (e.g., blood pressure, BMI), psychiatric symptoms, health-related quality of life, health behaviors (e.g., physical activity), and inpatient and outpatient use assessed at 6 and 12 months.

Impact: This study addresses VA HSR&D research priorities related to mental health and care of complex, chronic conditions, and is consistent with the priorities of the VHA's Office of Mental Health Services (Patient Care Services), 10NC, and the National Center for Health Promotion and Disease Prevention. Serious mental illness (SMI) is associated with significant disability, decreased quality of life, and a decreased life span. The VA is undergoing two major quality improvement initiatives: the Patient-Aligned Care Team (PACT), which involves enhanced access and continuity of care based on Chronic Care Model (CCM) principles, and dissemination of behavioral medicine programs. However, to date these programs have not been fully adapted to address gaps in quality or outcomes of care for Veterans with SMI. Findings from this RCT will inform ongoing VA transformational initiatives around systems redesign and behavioral medicine programs for Veterans with SMI and determine whether a customized CCM-behavioral medicine strategy is most effective in improving outcomes for this vulnerable group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of serious mental illness (schizophrenia, bipolar disorder, other psychosis, major depressive disorder, or other recurrent depression or affective disorder)
* Have at least one of the following risk factors for CVD (cardiovascular disease):

  * Body mass index (BMI) >28 or waist circumference of >35 (women) or >40 (men) inches OR
  * Self-reported diagnosis of hypertension ("high blood pressure"), dyslipidemia ("high cholesterol") or diabetes or high blood sugar OR
  * Documentation in the medical record of a diagnosis of or treatment for hypertension (defined as documented diagnosis or blood pressure of >140/90 on 2 occasions or prescription for an antihypertensive medication), dyslipidemia (documented diagnosis or LDL>160 or prescription for a lipid-lowering medication) or diabetes mellitus (documented diagnosis or HbA1C >7% or current prescription for oral hypoglycemic therapy)

Exclusion Criteria:

* Have unresolved substance intoxication or withdrawal, such as appearing to be intoxicated (e.g., incoherent, slurred speech), or experiencing withdrawal symptoms from substance abuse at the time of enrollment.
* Are unwilling or unable to provide informed consent or comply with study requirements at the time of enrollment (e.g., unable to complete forms or attend sessions due to substantial functional limitations).
* Active suicidal ideation at time of enrollment (focused interventions are more appropriate for this group)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M. Kilbourne, PhD MPH, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Kilbourne AM, Goodrich DE, Lai Z, Post EP, Schumacher K, Nord KM, Bramlet M, Chermack S, Bialy D, Bauer MS. Randomized controlled trial to assess reduction of cardiovascular disease risk in patients with bipolar disorder: the Self-Management Addressing Heart Risk Trial (SMAHRT). J Clin Psychiatry. 2013 Jul;74(7):e655-62. doi: 10.4088/JCP.12m08082. PMID 23945460
- [Result] O'Donnell AN, Williams M, Kilbourne AM. Overcoming roadblocks: current and emerging reimbursement strategies for integrated mental health services in primary care. J Gen Intern Med. 2013 Dec;28(12):1667-72. doi: 10.1007/s11606-013-2496-z. Epub 2013 Jun 4. PMID 23733375
- [Result] Goodrich DE, Kilbourne AM, Nord KM, Bauer MS. Mental health collaborative care and its role in primary care settings. Curr Psychiatry Rep. 2013 Aug;15(8):383. doi: 10.1007/s11920-013-0383-2. PMID 23881714
- [Result] Waxmonsky J, Kilbourne AM, Goodrich DE, Nord KM, Lai Z, Laird C, Clogston J, Kim HM, Miller C, Bauer MS. Enhanced fidelity to treatment for bipolar disorder: results from a randomized controlled implementation trial. Psychiatr Serv. 2014 Jan 1;65(1):81-90. doi: 10.1176/appi.ps.201300039. PMID 24129806
- [Result] Kilbourne AM, Bramlet M, Barbaresso MM, Nord KM, Goodrich DE, Lai Z, Post EP, Almirall D, Verchinina L, Duffy SA, Bauer MS. SMI life goals: description of a randomized trial of a collaborative care model to improve outcomes for persons with serious mental illness. Contemp Clin Trials. 2014 Sep;39(1):74-85. doi: 10.1016/j.cct.2014.07.007. Epub 2014 Jul 30. PMID 25083802
- [Derived] Kilbourne AM, Barbaresso MM, Lai Z, Nord KM, Bramlet M, Goodrich DE, Post EP, Almirall D, Bauer MS. Improving Physical Health in Patients With Chronic Mental Disorders: Twelve-Month Results From a Randomized Controlled Collaborative Care Trial. J Clin Psychiatry. 2017 Jan;78(1):129-137. doi: 10.4088/JCP.15m10301. PMID 27780336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 287 subjects completed baseline assessments, and 245 completed both baseline and 12-month follow-up assessments, and the 245 are included in final analyses, with 124 in the treatment (LGCC) group and 121 in the control (usual care) group.
Pre-assignment Details: 304 participants enrolled in the project, but only 287 completed baseline assessments, so those will be the participants included in the baseline analysis.
Groups:
- Arm 1 (Usual Care): Usual care will include standard mental health and medical care available in the VA clinics but with no active management by the LGCC health specialist.
- Arm 2 (Life Goals Collaborative Care): Life Goals Collaborative Care: LGCC consists of 1) 10 self-management sessions that cover personal goal-setting and mental health symptom management reinforced through healthy lifestyles; 2) medical care management that includes identification of patient medical risk factors, monitoring of patient symptoms and medical needs via a registry over time; and 3) support for provider guidelines and community linkages.
Period: Overall Study
Arm/Group | Arm 1 (Usual Care) | Arm 2 (Life Goals Collaborative Care)
Started | 146 | 141
Completed | 121 | 124
Not Completed | 25 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Usual Care) | Arm 2 (Life Goals Collaborative Care) | Total
Number analyzed (Participants) | 146 | 141 | 287
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 126 | 120 | 246
  >=65 years | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (11.0) | 55.3 (10.7) | 55.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 125 | 121 | 246
Region of Enrollment [Number; unit: participants]
  United States | 146 | 141 | 287

OUTCOME MEASURES:

1. Primary Outcome: Physical Health-related Quality of Life
Description: The outcome is measures by changes in the Veterans short form 12-item (VR-12) survey, which includes a physical and mental health component score (PCS and MCS, respectively). Each component score (PCS and MCS) has a range of 0-100, with a higher score on the PCS and MCS indicating better outcome, or better physical or mental health-related quality of life, respectively.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 (Usual Care) | Arm 2 (Life Goals Collaborative Care)
Number analyzed (Participants) | 121 | 124
units on a scale | 34.00 (11.49) | 33.61 (11.36)

2. Secondary Outcome: Improved Mental Health-related Quality of Life
Description: Change in SF-12 mental health scores from baseline to 12 months. The outcome is measures by changes in the Veterans short form 12-item (VR-12) survey, which includes a physical and mental health component score (PCS and MCS, respectively). Each component score (PCS and MCS) has a range of 0-100, with a higher score on the PCS and MCS indicating better outcome, or better physical or mental health-related quality of life, respectively.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1 (Usual Care): Usual care will include standard mental health and medical care available in the VA clinics but with no active management by the LGCC health specialist.
  .
Arm/Group | Arm 1 (Usual Care) | Arm 2 (Life Goals Collaborative Care)
Number analyzed (Participants) | 121 | 124
units on a scale | 36.36 (12.11) | 38.13 (12.41)

ADVERSE EVENTS:
Time Frame: During the course of the entire project, up to 1 year post-enrollment.
Arm/Group | Arm 1 (Usual Care) | Arm 2 (Life Goals Collaborative Care)
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/141
Other Adverse Events (participants affected / at risk) | 0/146 | 0/141

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No